CLINICAL TRIAL: NCT03889366
Title: Relative Bioavailability of NXP001 Compared to Emend® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuformix Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NXP001_01
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — Aprepitant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NXP001 Oral Capsule (Experimental)
  Interventions: Drug: Aprepitant 125 mg
- NXP001 Oral Suspension (Experimental)
  Interventions: Drug: Aprepitant 125 mg
- Emend® (Active Comparator)
  Interventions: Drug: Aprepitant 125 mg

INTERVENTIONS:
Drug: Aprepitant 125 mg — Single dose in the fasted state during treatment period 1,2 or 3

SUMMARY:
This study will compare the relative bioavailability of both an oral capsule formulation and an oral suspension formulation of NXP001 to Emend® in healthy male volunteers in the fasted state.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Body mass index (BMI) of 18.0 to 35.0 kg/m2 as assessed at screening
3. Must be willing and able to communicate and participate in the whole study
4. Must provide written informed consent
5. Must agree to use adhere to the contraception requirements of the study

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months prior to first dose
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. History of any drug or alcohol abuse in the past 2 years
4. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
5. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
6. Current users of e-cigarettes and nicotine replacement products and those who have smoked these products within the last 12 months
7. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
8. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
9. Confirmed positive drugs of abuse test result
10. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
11. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory, psychiatric or gastrointestinal (GI) disease as judged by the investigator
12. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
13. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
14. Donation or loss of greater than 400 mL of blood within the previous 3 months
15. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
16. Subjects who have taken any CYP3A4 inducers in the 30 days prior to IMP administration.
17. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC(0 to Infinity)) Following Single Dose Administration of NXP001 oral capsule, NXP001 oral suspension or Emend® in the fasted state | through 48 hours postdose

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) Following Single Dose Administration of NXP001 oral capsule, NXP001 oral suspension or Emend® in the fasted state | through 48 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Limited, Nottingham, United Kingdom